CLINICAL TRIAL: NCT06548321
Title: Benefits of Extracorporeal Shockwave Therapy to Reduce Spasticity in Stroke/CP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/735
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Cerebral
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracorporeal Shockwave Therapy (Experimental)
  Interventions: Diagnostic Test: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Diagnostic Test: Extracorporeal Shockwave Therapy — " The ESTW machine is turned on and the instrument, or shockwave gun, is pressed against the affected area. Rapid impulses are then delivered to the patient. Treatment typically lasts between 5 and 15 minutes. While this treatment can be uncomfortable for some, most do not experience any pain.
  Once treatment is completed, patients should do their best to physical activity… higher levels of energy Shockwaves into deeper tissue locations… ESWT therapies can help treat neurological disorders like multiple sclerosis and the effects of stroke.

SUMMARY:
This Study will help to explain us that ExtracorporealShockwave therapy can reduce spasticity in Stroke Patient,help them to restore their abilities and ROM.Therapy reduces dependency rate of patient.Also seen this therapy shows reduction in spasticity of CP child population.Improving the motor recovery.

DETAILED DESCRIPTION:
ESWT therapy increses molecular and immunological reactions,increase blood microcirculation and neurovascularization.It enhancing the neural proliferation of neural stem cell(NSC),which shows repair in brain function in CNS diseases.Extracorporeal shockwave can produce Nitric oxide in enzymatic and non enzymatic way which help, to reduce muscle spasm.Extracorporeal Shockwave reduce the exitibilty of motor neuron by vibratory stimulation of tendon and reduces tension.After 2 weeks ESWT muscle tension reduces increases range of motion reduces the pain.shock wave therapy appears to be effective in reducing spasticity levels irrespective of the age of the participants, the type of injury, and the tool used to measure the effect.ESWT change in motor neuron exitibilty & also associated with the spastic muscle.

ELIGIBILITY:
Inclusion Criteria:

* 3rd stage of Stroke

Exclusion Criteria:

* Non spastic CP,1st stage of Stroke,Spasticity caused by injury,Newborn

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale MAS | 12 Months
  The Ashworth Scale method of grading spasticity, working with Cerebral Palsy and Stroke patients. The original Ashworth scale was a 5 point numerical scale that graded spasticity from 0 to 4, with 0 being no resistance and 4 being a limb rigid in flexion or extension. In 1987, while performing a study to exam interrater reliability of manual tests of elbow flexor muscle spasticity, Bohannon and Smith modified the Ashworth scale by adding 1+ to the scale to increase sensitivity. Since its modification, the modified Ashworth scale (MAS), has been applied in clinical practice and research as a measure of spasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical setups Sargodha,Lahore,BWN, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No